CLINICAL TRIAL: NCT00324545
Title: Long-term Adherence and Cardiovascular Outcomes of a Randomized Controlled Trial of Medium-intensity Minimally-directive Counseling for Different Diets
Brief Title: Cardiovascular Outcomes Of Diet Counseling
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Camelot Foundation (Other)
Collaborators: GM Harrington, PhD (Unknown)
Responsible Party: Principal Investigator, RM Fleming, MD, PI, The Camelot Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000-1-1
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease; Obesity
Keywords: Obesity; Diets; Heart Disease; Randomized controlled trial; Ischemia.
MeSH Terms: conditions — Coronary Artery Disease; Obesity; Heart Diseases; Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: Medium-intensity Minimally-directive Counseling

SUMMARY:
(1) What effect does behavioral counseling for vegan, for low to moderate fat, and for lowered carbohydrate diets have on coronary blood flow? (2) What are the effects of different diet protocols when caloric intake and exercise are equalized? (3) Do people, so counseled, maintain their modified behaviors after they have completed their diet program? (4) How does targeting different diets affect secondary indices associated with heart disease such as weight, lipid, inflammatory, and thrombotic factors?

DETAILED DESCRIPTION:
Given the current epidemic of overweight and obesity on a global scale ("globesity") and the consequent world public health objective of reducing that obesity, it is evident as a practical matter that, the main line of attack must be through diet. The public health objective and the lack of information regarding the long-term public health effects of alternative weight-loss diets motivated this comparative study of the three major types of weight-loss diets and their long term effects on coronary blood flow. Secondary endpoints are inflammatory and other variables associated with heart disease and obesity.

Specifically we asked: (1) What effect does behavioral counseling for vegan, for low to moderate fat, and for lowered carbohydrate diets have on coronary blood flow? (2) What are the effects of different diet protocols when caloric intake and exercise are equalized? (3) Do people, so counseled, maintain their modified behaviors after they have completed their diet program? (4) How does targeting different diets affect secondary indices associated with heart disease such as weight, lipid, inflammatory, and thrombotic factors?

ELIGIBILITY:
Inclusion criteria: BMI greater than 30,

Exclusion criteria: pre-existing co-morbid diseases (documented heart disease, diabetes mellitus, cancer, hypertension, hepatic, renal or gastrointestinal disease), pregnancy or plans for pregnancy. Participants could not be smokers (cigarettes, cigars, pipes or chewing tobacco), take medications (prescription or over the counter medications with the exception of antibiotics), nor take vitamin or mineral supplements. Additionally, they could not currently be on a diet or have been on one during the last 6 months, or have food allergies that would influence food choices.

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2002-12-31 (Actual); Study Completion 2002-12-31

PRIMARY OUTCOMES:
coronary blood flow

SECONDARY OUTCOMES:
weight
BMI
LDLc
Total Cholesterol
HDLc
Triglycerides
Homocysteine
Fibrinogen
Lipoprotein (a)
VLDLc
TC/HDL
TG/HDL (Insulin Resistance)
CRP
IL-6
respiratory quotient

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Fleming, MD, Principal Investigator — Camelot Foundation; Gordon M Harrington, PhD, Principal Investigator — University of Northern Iowa
Locations (2):
- United States (2):
  - Keith Block, Chicago, Illinois
  - Richard M. Fleming, MD, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
Documents we are uploading onto Clinical Trials site.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We are uploading information onto the Clinical Trials site.
Access Criteria: Direct email request may be made to primary email.

REFERENCES:
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Bandura, A. (1986). Social foundations of thought and action: A social cognitive theory. xiii, 617.
- [Background] Bandura, A. (1997). Self-efficacy: The exercise of control. ix, 604.
- [Background] Barnard RJ. Effects of life-style modification on serum lipids. Arch Intern Med. 1991 Jul;151(7):1389-94. PMID 2064490
- [Background] Begg C, Cho M, Eastwood S, Horton R, Moher D, Olkin I, Pitkin R, Rennie D, Schulz KF, Simel D, Stroup DF. Improving the quality of reporting of randomized controlled trials. The CONSORT statement. JAMA. 1996 Aug 28;276(8):637-9. doi: 10.1001/jama.276.8.637. No abstract available. PMID 8773637
- [Background] Cantwell MM, Millen AE, Carroll R, Mittl BL, Hermansen S, Brinton LA, Potischman N. A debriefing session with a nutritionist can improve dietary assessment using food diaries. J Nutr. 2006 Feb;136(2):440-5. doi: 10.1093/jn/136.2.440. PMID 16424125
- [Background] Dansinger ML, Gleason JA, Griffith JL, Selker HP, Schaefer EJ. Comparison of the Atkins, Ornish, Weight Watchers, and Zone diets for weight loss and heart disease risk reduction: a randomized trial. JAMA. 2005 Jan 5;293(1):43-53. doi: 10.1001/jama.293.1.43. PMID 15632335
- [Background] DAVIS CM. Self regulation of diet in childhood. Health Educ J (Los Angel). 1947 Jan;5:37-40. doi: 10.1177/001789694700500110. No abstract available. PMID 20247154
- [Background] Fleming, R. M. (1999). The pathogenesis of vascular disease. In J. Chang (Ed.), The Textbook of Angiology (pp. 787-798). New York: Springer-Verlag.
- [Background] Fleming RM. The effect of high-protein diets on coronary blood flow. Angiology. 2000 Oct;51(10):817-26. doi: 10.1177/000331970005101003. PMID 11108325
- [Background] Fleming RM. Reversing heart disease in the new millennium--the Fleming unified theory. Angiology. 2000 Aug;51(8):617-29. PMID 10959514
- [Background] Fleming RM. The effect of high-, moderate-, and low-fat diets on weight loss and cardiovascular disease risk factors. Prev Cardiol. 2002 Summer;5(3):110-8. doi: 10.1111/j.1520-037x.2002.01231.x. PMID 12091753
- [Background] Fleming RM, Ketchum K, Fleming DM, Gaede R. Treating hyperlipidemia in the elderly. Angiology. 1995 Dec;46(12):1075-83. doi: 10.1177/000331979504601202. PMID 7495312
- [Background] Fleming RM, Ketchum K, Fleming DM, Gaede R. Assessing the independent effect of dietary counseling and hypolipidemic medications on serum lipids. Angiology. 1996 Sep;47(9):831-40. doi: 10.1177/000331979604700901. PMID 8810649